CLINICAL TRIAL: NCT07332494
Title: Digital Remote Management for Care and Continuous Optimization Versus Usual Care in Patients With Coronary Heart Disease (DigiCare-CHD)
Acronym: DigiCare-CHD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Chang sheng Ma, Director of cardiology department, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KS2025290
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Coronary Heart Disease; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care Group (No Intervention): Patients receive standard post-PCI management, including guideline-directed medical therapy (GDMT) and routine outpatient follow-up visits at 1, 3, 6, 9, and 12 months.
- Digital Remote Management Group (Experimental): 1-year intervention:
  1. BP Management: Protocol-driven self-monitoring frequencies. The system triggers alerts for BP >130/80 mmHg and generates automated suggestions for medication titration, subject to physician approval.
  2. Lipid Management: Automated reminders for laboratory testing. Optical Character Recognition (OCR) technology extracts data from lab reports. If LDL-C ≥1.4 mmol/L, the system proposes regimen intensification for physician review.
  3. Exercise Management:Target of ≥6000 steps/day. Data is synchronized via wearables or smartphones. Inactivity triggers automated behavioral feedback.
  4. Medication Management: Daily app-based reminders and digital "check-ins." Non-adherence triggers automated alerts followed by human intervention if persistent.
  5. Symptom Monitoring: Patient-reported outcomes (e.g., chest pain/dyspnea) via the App, with automated triage for risk stratification.
  6. Health Education: Push delivery of targeted secondary prevention educational materials.
  Interventions: Other: Digital Remote Management Group

INTERVENTIONS:
Other: Digital Remote Management Group — 1-year intervention
  1. BP Management: Protocol-driven self-monitoring frequencies. The system triggers alerts for BP >130/80 mmHg and generates automated suggestions for medication titration, subject to physician approval.
  2. Lipid Management: Automated reminders for laboratory testing. Optical Character Recognition (OCR) technology extracts data from lab reports. If LDL-C ≥1.4 mmol/L, the system proposes regimen intensification for physician review.
  3. Exercise Management:Target of ≥6000 steps/day. Data is synchronized via wearables or smartphones. Inactivity triggers automated behavioral feedback.
  4. Medication Management: Daily app-based reminders and digital "check-ins." Non-adherence triggers automated alerts followed by human intervention if persistent.
  5. Symptom Monitoring: Patient-reported outcomes (e.g., chest pain/dyspnea) via the App, with automated triage for risk stratification.
  6. Health Education: Push delivery of targeted secondary prevention educational materials.
  Arms: Digital Remote Management Group

SUMMARY:
The DigiCare-CHD study is an investigator-initiated, multicenter, open-label, parallel-group randomized controlled trial. It aims to evaluated the efficacy of a smartphone-based digital remote management platform compared to usual care in achieving dual goal attainment of blood pressure and LDL-cholesterol levels in patients with coronary heart disease following percutaneous coronary intervention.

DETAILED DESCRIPTION:
"Coronary heart disease (CHD) remains a leading cause of global mortality. While percutaneous coronary intervention (PCI) significantly improves acute survival, patients continue to face substantial residual cardiovascular risk driven by the progression of systemic atherosclerosis. Rigorous management of blood pressure (BP) and low-density lipoprotein cholesterol (LDL-C) is imperative for secondary prevention. However, achieving simultaneous targets (BP < 130/80 mmHg and LDL-C < 1.4 mmol/L) in real-world practice is challenging due to clinical inertia and suboptimal patient adherence. Traditional outpatient follow-up is often fragmented and reactive, failing to provide the continuous monitoring required for optimal risk factor control.

The DigiCare-CHD trial serves as a prospective, multicenter, open-label randomized controlled trial designed to enroll 792 patients who have successfully undergone PCI for acute or chronic coronary syndromes. Participants will be randomized 1:1 to either the Digital Remote Management group or the Usual Care group, with a follow-up period of 12 months.

Patients in the intervention arm will utilize a digital remote management platform. This system integrates home monitoring to track BP, lipid profiles, and physical activity. Key features include AI-driven alerts for abnormal values, automated decision support for medication titration (verified by physicians), and targeted health education. The primary endpoint is the rate of dual goal attainment for BP and LDL-C at 12 months. DigiCare-CHD aims to establish a proactive, closed-loop management strategy to effectively reduce residual cardiovascular risk and improve long-term prognosis in the post-PCI population."

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Diagnosis of Acute Coronary Syndrome (ACS) or Chronic Coronary Syndrome (CCS)
3. Status post-successful percutaneous coronary intervention (PCI).
4. Possession of a smartphone and ability to operate the application (independently or with caregiver assistance).
5. Provision of written informed consent.

Exclusion Criteria:

1. Heart Failure: NYHA Class III-IV or LVEF < 40%.
2. Severe hepatic dysfunction (ALT/AST ≥3xULN or Total Bilirubin >1.5 mg/dl)
3. Severe renal dysfunction (eGFR < 30 ml/min/1.73m² or requiring dialysis)
4. Uncontrolled hypothyroidism (TSH >1.5xULN or >10 mIU/L, or unstable dosage within 6 weeks)
5. Life expectancy < 1 year due to non-cardiovascular comorbidities
6. Severe sensory (hearing/vision) or cognitive impairment precluding device use
7. Conditions affecting adherence (e.g., substance use disorder, history of alcohol abuse)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 792 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Dual Goal Attainment for Blood Pressure and Lipids | 12 months after randomization
  Defined as the proportion of patients achieving both SBP < 130 mmHg and DBP < 80 mmHg and LDL-C < 1.4 mmol/L.

SECONDARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) | Baseline and 12 Months
Exercise Compliance Rate | 12 Months
  Proportion of patients maintaining an average of ≥6000 steps/day.
Medication Adherence | 12 Months
  MARS-10 scale
Smoking Cessation Rate | 12 Months
  Self-reported complete abstinence from smoking among baseline smokers
Quality of Life（EQ-5D-5L） | 12 Months
  EQ-5D-5L
Major Adverse Cardiovascular Events (MACE) Composite of all-cause death, myocardial infarction, malignant arrhythmia, or hospitalization for heart failure. | 12 Months

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - 13810720787, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing, China, Beijing
  - The First Affiliated Hospital of Dalian Medical University, Dalian, China, Dalian
  - The First Hospital of Jilin University, Changchun, China, Jilin

IPD SHARING:
Plan to Share IPD: No